CLINICAL TRIAL: NCT06115980
Title: First in Man, Open-label, Multi Center Safety and Preliminary Performance of Xtrac O.S. System for Lead Extraction.
Brief Title: Safety and Preliminary Performance of Xtrac O.S. System for Lead Extraction.
Acronym: XTR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xtrac O.S. (Industry)
Collaborators: KCRI (Other); Scopus Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XTR-01-0322
Record Dates: First submitted 2023-07-20; First posted 2023-11-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized, feasibility, prospective, interventional clinical trial of lead extraction.
  The Xtrac O.S. system is intended for transvenous removal of pacing or defibrillator leads, having an inner lumen, through a superior approach.
  A total of 10 patients, who are scheduled for lead extraction, will be recruited in order to ensure a total of at least 10 patients finishing the study procedures and follow up.
  The decision upon lead extraction will be based upon the applicable Heart Rhythm Society guidelines or European Heart Rhythm Association (EHRA).
  Each enrolled patient will undergo a pre procedural evaluation to enable planning of the extraction procedure. The evaluation includes an assessment of the CIED components to be removed, dwell time, anatomic course on radiography and patient characteristics that may require management prior to extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 - An open label study (Experimental): This is an open label, non-randomized, feasibility, prospective, interventional clinical trial of lead extraction. The Xtrac O.S. system is intended for transvenous removal of pacing or defibrillator leads, having an inner lumen, through a superior approach.
  A total of 15 patients, who are scheduled for lead extraction, will be recruited in order to ensure a total of at least 10 patients finishing the study procedures and follow up.
  Interventions: Device: lead extraction (Xtrac O.S. system)

INTERVENTIONS:
Device: lead extraction (Xtrac O.S. system) — This is an open label, non-randomized, feasibility, prospective, interventional clinical trial of lead extraction. The Xtrac O.S. system is intended for transvenous removal of pacing or defibrillator leads, having an inner lumen, through a superior approach.
  The decision upon lead extraction will be based upon the applicable Heart Rhythm Society guidelines or European Heart Rhythm Association (EHRA).
  Each enrolled patient will undergo a pre procedural evaluation to enable planning of the extraction procedure. The evaluation includes an assessment of the CIED components to be removed, dwell time, anatomic course on radiography and patient characteristics that may require management prior to extraction.
  A multidisciplinary team evaluation involving cardiac surgery, electrophysiologist, and cardiac anesthesiology should allow for a rapid and successful response to major complications

SUMMARY:
This is an open label, interventional, feasibility, prospective, multicenter, clinical trial of lead extraction. The Xtrac O.S. system is intended for transvenous removal of pacing or defibrillator leads, having an inner lumen, through a superior approach.

A total of 15 patients, who are scheduled for CIED lead extraction, will be recruited in order to ensure a total of at least 10 patients finishing the study procedures and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Men or Female patients, 18-85 years old.
2. Patients must understand the procedures and methods of this study and be willing to sign the informed consent form and to complete the trial in strict accordance with clinical trial protocol.
3. Scheduled for a CIED lead extraction upon current guidelines.
4. Lead implant duration more than 1 year and less than 5 years.
5. Patient must be SARS-CoV-2 negative and without Covid-19 signs and symptoms, prior to enrollment.
6. Patients are classified as ASA II/III.
7. Leads with external diameter of 7Fr-9Fr.

Exclusion Criteria:

1. Patient age > 85 years old.
2. Hemodynamic instability.
3. Class IV NYHA heart failure.
4. Contrast allergy.
5. Patients felt to be high risk due to degree of acute illness or systemic comorbidities.
6. Patients who are placed on a heparin bridge, and are felt to be high risk for even brief discontinuation of anticoagulation
7. Pregnant or lactating.
8. Participating in another clinical study.

Eligibility will be determined by the PI and investigators based on the exclusion/inclusion criteria, current medical status and evaluation of the procedure risks mitigation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety related to the lead extraction procedure, or the extraction tool | 0 to 30 days post-lead extraction
  To collect and evaluate device- and procedure-related adverse events.

SECONDARY OUTCOMES:
To assess the ease of use, duration of the procedure and the physician satisfaction by questions by a Likert scale | During procedure
  Using Likert scale (1 - Poor; 2 - Fair; 3 - Good; 4 - Excellent)
To evaluate the rate of complete procedural success of removal leads implanted for more than 1and up to 5 years | Acute setting (during the surgical procedure)
  Complete procedural success is the removal of the targeted lead and all lead material from the vascular space, with the absence of permanently disabling complications or procedure-related death
To evaluate the rate of clinical procedural success | Acute setting (during the surgical procedure)
  Clinical procedural success is the removal of all targeted leads and all lead material from the vascular space, or retention of a small portion of the lead (fragment that is 4 cm or smaller) that does not negatively impact the outcome goals of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel